CLINICAL TRIAL: NCT01554124
Title: Pharmacokinetics and Safety of Meropenem in Infants Below 90 Days of Age (Inclusive) With Probable and Confirmed Meningitis: A European Multicenter Phase I-II Trial
Brief Title: Pharmacokinetics and Safety of Meropenem in Infants Below 90 Days of Age With Probable and Confirmed Meningitis
Acronym: NeoMero-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001521-25
Record Dates: First submitted 2012-02-27; First posted 2012-03-14 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Meningitis
Keywords: Meningitis; Neonates; Meropenem
MeSH Terms: conditions — Meningitis | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Meropenem (Experimental): Infants will received Meropenem 40 mg/kg every 8 hours (every 12 hours in the youngest age group: < 32 weeks GA and < 2 weeks postnatal age).
  Treatment duration = 21 ± 7 days
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — 40 mg/kg every 8 hours (every 12 hours in the youngest age group: < 32 weeks GA and < 2 weeks postnatal age).
  Treatment duration = 21 ± 7 days
  Other Names: Meropenem trihydrate

SUMMARY:
This phase I-II multicenter international trial is designed to study the pharmacokinetics of meropenem and to characterize the safety profile of meropenem in the treatment of infants ≤ 90 days of postnatal age with probable or confirmed bacterial meningitis.

DETAILED DESCRIPTION:
The primary objective will be to study the pharmacokinetics (plasma and cerebrospinal fluid) of meropenem in infants ≤ 90 days of postnatal age with probable or confirmed bacterial meningitis and to characterize the safety profile of meropenem in the treatment of infants ≤ 90 days of postnatal age with probable or confirmed bacterial meningitis.

The secondary objectives are :

* To describe the efficacy of meropenem on day 3, at end of allocated treatment (EOAT), at test of cure (TOC) and at follow up (FU).
* To evaluate survival at FU
* To evaluate further episodes of meningitis (relapse or new infection) occurring between TOC and FU visits
* To define the organisms causing neonatal meningitis
* To describe the antibacterial susceptibility of meningitis-causing organisms and to describe the clinical and microbiological response according to this
* To evaluate mucosal colonization by resistant organisms before and after treatment with meropenem
* To evaluate bacterial eradication
* To evaluate functional genetic parameters that may affect response to therapy

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the parents/carers
* Chronological age below 90 days inclusive
* The presence of:

  * clinical signs consistent with BM (hyperthermia or hypothermia or temperature instability PLUS 1 or more neurological findings among coma, seizures, neck stiffness, apnoea, bulging fontanelle),
  * OR CSF pleocytosis (≥ 20 cells/mm3)
  * OR a positive Gram stain of CSF.

Exclusion Criteria:

* Presence of a CSF device
* Proven viral or fungal meningitis
* Severe congenital malformations if the infant is not to expect to survive for more than 3 months
* Other situations where the treating physician considers a different empiric antibiotic regimen necessary
* Known intolerance or contraindication to the study medication
* Participation in any other clinical study of an investigational medicinal product
* Renal failure and requirement of haemofiltration or peritoneal dialysis
* Meningitis with an organism known to be resistant to meropenem

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Meropenem (plasma and CSF) in infants ≤ 90 days of age diagnosed with probable and confirmed bacterial meningitis. | 3-4 days
  Pharmacokinetic analyses (AUC) will be carried out on the infants who received at least one dose of meropenem after inclusion in NeoMero-2.
  The final model will be used for dosing simulations to give final dose recommendations.
Nature, frequency and numbers of all adverse events under meropenem. | Up to 48 days
  Adverse events will also be summarised according to the need of a specific medical intervention or not. Analyses by time period will also be shown (from D0 to TOC visit and from TOC visit to follow-up).

SECONDARY OUTCOMES:
Percentage of patients with a favourable outcome defined at Test of Cure visit (TOC). | An expected average of 21 days
  Patients with a favourable outcome defined at Test of Cure visit (TOC) 2 days after EOAT is met as an infant fulfilling the following criteria: Alive with clinical and bacteriological resolution of the abnormalities that defined BM at entry and no occurrence of any new clinical or laboratory abnormalities requiring a new course of antibiotic therapy and no modification of the initial meropenem therapy (for more than 24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Paul HEATH, Principal Investigator — Paediatric Infectious Diseases St Georges, University of London; Jean-Pierre ABOULKER, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- HEATH, Paul, London, Cranmer Terrace, United Kingdom

REFERENCES:
- See also: Site dedicated to the NeoMero studies — http://www.neomero.org